CLINICAL TRIAL: NCT01596257
Title: Randomized Phase II Trial of Bulk Versus Fractionated Stem Cell Infusions in Patients With Hematologic Malignancies Undergoing Stem Cell Transplantation
Brief Title: Bulk Versus Fractionated Stem Cell Infusions in Patients With Hematologic Malignancies Undergoing Stem Cell Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-016
Record Dates: First submitted 2012-05-09; First posted 2012-05-10 (Estimated); Results first posted 2022-12-29 (Actual); Last update posted 2022-12-29 (Actual); Status verified 2021-08

CONDITIONS: Leukemia
Keywords: CliniMACS-CD34 Reagent System; Acute Leukemia; Myelodysplastic syndrome; Non Hodgkins Lymphoma; Hodgkins Disease; Multiple Myeloma; 12-016
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Lymphoma, Non-Hodgkin; Hodgkin Disease; Multiple Myeloma

ARMS (2):
- bulk SCT (Active Comparator): Patients receive reduced intensity or myeloablative conditioning regimen, GVHD prophylaxis, and undergo T cell depleted or no T cell depleted allogeneic SCT on day 0. After completion of study treatment, patients are followed up every 6-8 weeks for up to 24 months
  Interventions: Procedure: allogeneic hematopoietic stem cell transplantation; Device: CliniMACS
- fractionated SCT (Experimental): Patients receive reduced intensity or myeloablative conditioning regimen, GVHD prophylaxis, and undergo T cell depleted or no T cell depleted allogeneic SCT on days 0, 2, 4, and 6. After completion of study treatment, patients are followed up every 6-8 weeks for up to 24 months
  Interventions: Procedure: allogeneic hematopoietic stem cell transplantation; Device: CliniMACS

INTERVENTIONS:
Procedure: allogeneic hematopoietic stem cell transplantation — Undergo allogeneic hematopoietic stem cell transplant
Device: CliniMACS

SUMMARY:
The purpose of this study is to find out if getting a blood stem cell transplant with donor stem cells given over several days is better than getting a blood stem cell transplant with donor stem cells given over 1 day. We want to find out which procedure over will result in improved recovery of blood and immune function after transplant. When donor stem cells are given over various days in mice, the blood and immune system recovery is quicker.

DETAILED DESCRIPTION:
This is a complex study that involves various interventions, Intervention #1: Donor Initial Stem Cell Collection; Intervention #2: Stem Cell Product Initial Processing Orders; Intervention #3 Patient Admission and Transplantation; Intervention #4: Stem cell infusion; Intervention #5: Post infusion follow up; Intervention #6: Off Study Patient and Donor Evaluation.

Patients whose donor fails to collect the appropriate number of cells will receive all their cells as a bulk infusion. These patients will continue to receive a transplant on protocol but will be replaced until both arms have reached the target accrual.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are considered candidates for an allogeneic stem cell transplantation as treatment for any of the following hematologic disorders:
* Acute Leukemia
* Myelodysplastic syndrome
* Other myeloproliferative disorder (i.e. myelofibrosis, chronic myelomonocytic leukemia, or chronic myelogenous leukemia)
* Non Hodgkins Lymphoma
* Hodgkins Disease
* Multiple Myeloma
* Age includes from birth to < 75 years old.
* Patients must have a Karnofsky (adult) or Lansky (pediatric) Performance Status > 70%
* Patients must have adequate organ function measured by:
* Cardiac: asymptomatic or if symptomatic then LVEF at rest must be > 40%
* Hepatic: < 5x ULN ALT and < 1.5 total serum bilirubin, unless there is congenital benign hyperbilirubinemia.
* Renal: serum creatinine <1.5 mg/dl or if serum creatinine is outside the normal range, then CrCl > 40 ml/min (measured or calculated/estimated)
* Pulmonary: asymptomatic or if symptomatic, DLCO > 40% of predicted (corrected for hemoglobin).

Exclusion Criteria:

* Female patients who are pregnant or breast-feeding.
* Active viral, bacterial or fungal infection
* Patient seropositive for HIV-I/II; HTLV -I/II
* Presence of leukemia in the CNS
* Candidate for a protocol of higher priority. For the purpose of this study, the following protocols will be considered of higher priority: 10-051

Donor Inclusion Criteria:

* HLA compatible related or unrelated donor, (i.e. a fully matched unmanipulated grafts or 1-2 HLA allele disparate donor for CD34 selected grafts).
* Meets criteria outlined in the FACT-approved SOP for "DONOR EVALUATION AND SELECTION FOR ALLOGENEIC TRANSPLANTATION" in the Blood and Marrow Transplant Program Manual, document E-1 see http://mskweb5.mskcc.org/intranet/html/80312.cfm
* Donor must have adequate peripheral venous catheter access for leukapheresis or must agree to placement of a central catheter.
* Wt >25kg

Donor Exclusion Criteria:

* Evidence of active infection (including urinary tract infection, or upper respiratory tract Infection) or viral hepatitis exposure (on screening), unless only HBS Ab+ and HBV DNA negative.
* Medical or physical reason which makes the donor unlikely to tolerate or cooperate with growth factor therapy and leukapheresis.
* Factors which place the donor at increased risk for complications from leukapheresis or GCSF therapy (e.g., autoimmune disease, sickle cell trait, symptomatic coronary artery disease requiring therapy).
* Pregnancy (positive serum or urine β-HCG) or breastfeeding. Women of childbearing age must avoid becoming pregnant while on the study

Max Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2012-05-05 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Giralt, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study goal was to explore fractionated HPC infusion in humans in a setting of commonly used conditioning regimens. The design included stratification of randomization by transplant type. Additional stratification would have increased the accrual target for statistical power, prolonging enrollment. In our publication reporting results of this trial (Tamari et al. JTCT 2021) we provide data stratified by treatment arm and transplant type for secondary endpoints for easier interpretation.
Groups:
- Bulk Stem Cell Transplantation/SCT: Patients receive reduced intensity or myeloablative conditioning regimen, GVHD prophylaxis, and undergo T cell depleted or no T cell depleted allogeneic SCT on day 0. After completion of study treatment, patients are followed up every 6-8 weeks for up to 24 months
  allogeneic hematopoietic stem cell transplantation: Undergo allogeneic hematopoietic stem cell transplant
  CliniMACS
- Fractionated Stem Cell Transplantation/SCT: Patients receive reduced intensity or myeloablative conditioning regimen, GVHD prophylaxis, and undergo T cell depleted or no T cell depleted allogeneic SCT on days 0, 2, 4, and 6. After completion of study treatment, patients are followed up every 6-8 weeks for up to 24 months
  allogeneic hematopoietic stem cell transplantation: Undergo allogeneic hematopoietic stem cell transplant
  CliniMACS
Period: Overall Study
Arm/Group | Bulk Stem Cell Transplantation/SCT | Fractionated Stem Cell Transplantation/SCT
Started | 61 | 55
Completed | 38 | 36
Not Completed | 23 | 19
Not completed — Inadequate Collection | 23 | 19

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bulk Stem Cell Transplantation/SCT | Fractionated Stem Cell Transplantation/SCT | Total
Number analyzed (Participants) | 61 | 55 | 116
Age, Continuous [Median (Full Range); unit: years] | 59 [13 to 70] | 59 [24 to 73] | 59 [13 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 19 | 49
  Male | 31 | 36 | 67
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 0 | 5
  Not Hispanic or Latino | 56 | 55 | 111
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 5 | 5
  White | 51 | 48 | 99
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 6 | 2 | 8
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 61 | 55 | 116

OUTCOME MEASURES:

1. Primary Outcome: Median Time to Engraftment of Neutrophils
Description: Determine the effects of fractionated vs. bulk stem cell infusions on neutrophil recovery as defined by number of days with an absolute neutrophil count of less than 500 neutrophils per micro liter and time to an absolute neutrophil count (ANC) of 500. Determing the median time to ANC of >/= 0.5 x 10^9/L
Time Frame: Up to 100 weeks
Measure: Median (Full Range); unit: days
Arm/Group | Bulk Stem Cell Transplantation/SCT | Fractionated Stem Cell Transplantation/SCT
Number analyzed (Participants) | 38 | 36
days | 11 [9 to 22] | 11 [9 to 22]

2. Secondary Outcome: Number of Participants Assessed for Toxicities
Description: Participants will be assessed for toxicities with the NCI-Common Terminology for Adverse Events (CTCAE), version 4.0.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Groups:
- Bulk SCT: Patients receive reduced intensity or myeloablative conditioning regimen, GVHD prophylaxis, and undergo T cell depleted or no T cell depleted allogeneic SCT on day 0. After completion of study treatment, patients are followed up every 6-8 weeks for up to 24 months
  allogeneic hematopoietic stem cell transplantation: Undergo allogeneic hematopoietic stem cell transplant
  CliniMACS
- Fractionated SCT: Patients receive reduced intensity or myeloablative conditioning regimen, GVHD prophylaxis, and undergo T cell depleted or no T cell depleted allogeneic SCT on days 0, 2, 4, and 6. After completion of study treatment, patients are followed up every 6-8 weeks for up to 24 months
  allogeneic hematopoietic stem cell transplantation: Undergo allogeneic hematopoietic stem cell transplant
  CliniMACS
Arm/Group | Bulk SCT | Fractionated SCT
Number analyzed (Participants) | 61 | 55
Participants
  Participants who experienced toxicities | 38 | 36
  Participants who did not experience toxicities | 23 | 19

3. Secondary Outcome: Median Time to Platelet Engraftment
Description: The area under the hematopoietic recovery curve for the factors: ALC, CD4, CD8, and platelet count. The area under the curve will be computed based on recordings at days 30, 60, 100, 180, 365. Determine days to platelet engraftment by platelet count.
Time Frame: Up to 365 days
Measure: Median (Full Range); unit: days
Arm/Group | Bulk SCT | Fractionated SCT
Number analyzed (Participants) | 38 | 36
days | 18 [9 to 112] | 18 [4 to 47]

4. Secondary Outcome: Overall Survival
Description: Percentage of participants alive at 24 months
Time Frame: 24 months
Measure: Number; unit: % of participants alive
Arm/Group | Bulk SCT | Fractionated SCT
Number analyzed (Participants) | 38 | 36
% of participants alive | 60 | 62

5. Secondary Outcome: Hematopoietic Function on Day 30
Description: Determine the difference of CD4+ lymphocyte recovery between the two arms on day 30
Time Frame: 30 days
Measure: Median (Full Range); unit: cells/mm^3
Arm/Group | Bulk SCT | Fractionated SCT
Number analyzed (Participants) | 38 | 36
cells/mm^3 | 0 [0 to 1473] | 6 [0 to 678]

6. Secondary Outcome: Hematopoietic Function on Day 180
Description: Determine the difference of CD4+ lymphocyte recovery between the two arms on day 180
Time Frame: 180 days
Measure: Median (Full Range); unit: cells/mm^3
Arm/Group | Bulk SCT | Fractionated SCT
Number analyzed (Participants) | 38 | 36
cells/mm^3 | 179 [0 to 799] | 111 [0 to 4180]

7. Secondary Outcome: Hematopoietic Function on Day 360
Description: Determine the difference of CD4+ lymphocyte recovery between the two arms on day 360
Time Frame: 360 days
Measure: Median (Full Range); unit: cells/mm^3
Arm/Group | Bulk SCT | Fractionated SCT
Number analyzed (Participants) | 38 | 36
cells/mm^3 | 294 [0 to 1076] | 280 [27 to 928]

ADVERSE EVENTS:
Time Frame: 2 years
Description: Data was pre-specified to be collected for aggregate Bulk SCT and Fractionated SCT interventions and not per transplant type stratification. Adverse Events were not collected based on transplant type stratification
Arm/Group | Bulk Stem Cell Transplantation/SCT | Fractionated Stem Cell Transplantation/SCT
All-Cause Mortality (participants affected / at risk) | 26/61 | 23/55
Serious Adverse Events (participants affected / at risk) | 21/61 | 12/55
Other Adverse Events (participants affected / at risk) | 38/61 | 36/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bulk Stem Cell Transplantation/SCT (N=61) | Fractionated Stem Cell Transplantation/SCT (N=55)
Anemia (Blood and lymphatic system disorders) | 1 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1
Blood and lymphatic system disorders - Other, spec (Blood and lymphatic system disorders) | 0 | 1
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Catheter related infection (Infections and infestations) | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0
Confusion (Psychiatric disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Cystitis noninfective (Renal and urinary disorders) | 0 | 1
Death NOS (General disorders) | 3 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 3 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Endocrine disorders - Other, specify (Endocrine disorders) | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 0
Fever (General disorders) | 3 | 0
Fracture (Injury, poisoning and procedural complications) | 1 | 0
Heart failure (Cardiac disorders) | 0 | 1
Hematuria (Renal and urinary disorders) | 1 | 0
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 1 | 1
Hypotension (Vascular disorders) | 1 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 7 | 2
Infections and infestations - Other, specify (Infections and infestations) | 3 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1
Intracranial hemorrhage (Nervous system disorders) | 1 | 1
Lethargy (Nervous system disorders) | 0 | 1
Lung infection (Infections and infestations) | 7 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 2
Neutrophil count decreased (Investigations) | 0 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Platelet count decreased (Investigations) | 1 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Seizure (Nervous system disorders) | 1 | 0
Sepsis (Infections and infestations) | 1 | 1
Syncope (Nervous system disorders) | 0 | 1
Urinary frequency (Psychiatric disorders) | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0
Urinary urgency (Renal and urinary disorders) | 1 | 0
Vasculitis (Vascular disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 2
White blood cell decreased (Investigations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bulk Stem Cell Transplantation/SCT (N=61) | Fractionated Stem Cell Transplantation/SCT (N=55)
Febrile Neutropenia (Blood and lymphatic system disorders) | 20 | 23
Infections and infestations - Other, specify (Infections and infestations) | 23 | 12
Mucositis oral (Gastrointestinal disorders) | 30 | 17
Hypertension (Vascular disorders) | 3 | 7
Hypotension (Vascular disorders) | 11 | 7
Colitis (Gastrointestinal disorders) | 7 | 0
Skin & subcutaneous tissue disorders Other, spec (Skin and subcutaneous tissue disorders) | 0 | 3
Abdominal pain (Gastrointestinal disorders) | 0 | 6
Alanine aminotransferase increased (Investigations) | 12 | 11
Alkaline phosphatase increased (Investigations) | 3 | 3
Allergic reaction (Immune system disorders) | 3 | 3
Anorexia (Metabolism and nutrition disorders) | 18 | 13
Anxiety (Psychiatric disorders) | 4 | 0
Aspartate aminotransferase increased (Investigations) | 4 | 6
Blood bilirubin increased (Investigations) | 6 | 3
Catheter related infection (Infections and infestations) | 10 | 8
Cholecystitis (Hepatobiliary disorders) | 3 | 0
Confusion (Psychiatric disorders) | 3 | 0
Dehydration (Metabolism and nutrition disorders) | 5 | 0
Diarrhea (Gastrointestinal disorders) | 19 | 19
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 | 7
Esophagitis (Gastrointestinal disorders) | 4 | 3
Fatigue (General disorders) | 9 | 7
Headache (Nervous system disorders) | 4 | 3
Hyperglycemia (Metabolism and nutrition disorders) | 24 | 13
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 11 | 7
Infusion related reaction (Injury, poisoning and procedural complications) | 4 | 0
Lung infection (Infections and infestations) | 19 | 7
Nausea (Gastrointestinal disorders) | 18 | 15
Pain (General disorders) | 0 | 5
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 14 | 11
Sinus tachycardia (Cardiac disorders) | 4 | 0
Syncope (Nervous system disorders) | 4 | 0
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 3 | 0
Vomiting (Gastrointestinal disorders) | 8 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-30): https://cdn.clinicaltrials.gov/large-docs/57/NCT01596257/Prot_SAP_000.pdf